CLINICAL TRIAL: NCT04389164
Title: A Multicenter, Randomized, Controlled Clinical Trial of Tissue-engineered Skin Grafts With Autologous Scar Dermal Scaffolds for the Repair of Hypertrophic Scars
Brief Title: Tissue-engineered Skin Graft Repair of Autologous Scar Dermal Scaffolds
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhu Jiayuan, Professor, associate chief physician, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018002
Record Dates: First submitted 2020-04-29; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Scar
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tissue engineering method (Experimental): The thickness of scar tissue in the middle of the dermis is removed by a roller cutter with a thickness of about 0.01 -- 0.02mm. After cleaning, the dermis can be used for punching and mesh drawing in the dermal rolling machine.Autologous epidermal basal cell suspension was prepared according to the description of autologous epidermal basal cell extraction box.The size of the remaining skin should be the same as the wound surface. After washing with normal saline, the wet yarn should be wrapped for later use.The autogenous scar dermal scaffold was prepared and transplanted onto the wound surface. The autoepidermal basal cells prepared were sprayed or coated between the mesh and the dermal scaffold. Autologous skin slices were transplanted onto the wound surface and fixed with pressure bandaging.
  Interventions: Procedure: Tissue-engineered skin grafts of autologous scar dermal scaffolds
- Conventional therapy (Active Comparator): Autologous skin was grafted onto the wound surface and fixed with pressure bandage
  Interventions: Procedure: Tissue-engineered skin grafts of autologous scar dermal scaffolds

INTERVENTIONS:
Procedure: Tissue-engineered skin grafts of autologous scar dermal scaffolds — 1. scar excision. The thickness of scar tissue in the middle of scar is removed with a roller cutter and the thickness is about 0.01 -- 0.02mm.
  2. take autologous skin slices of the patient with an electric skin knife, cut out a small piece of skin, and prepare autologous epidermal basal cell suspension for use;The rest of the skin should be the same size as the wound.
  3. the prepared autogenous scar dermal stent was grafted onto the scar resection wound surface, and the prepared autoepidermal basal cells were sprayed between the mesh and on the dermal stent, and autologous skin slices were grafted onto the wound surface and fixed with pressure bandaging;
  4. after the operation, the outer dressing should be changed regularly according to the conventional treatment, and the wound surface condition should be observed and recorded according to the experimental scheme.

SUMMARY:
Hypertrophic scar is an inevitable outcome of wound repair. It affects the appearance and some scar contracture often leads to joint dysfunction.Patients have low quality of life, long treatment cycle, heavy social burden and high medical costs.Skin grafting is currently the gold standard for scar repair.However, there are often insufficient skin sources, easy to scar recurrence, lack of skin accessory organs.The application of composite skin graft can reduce the recurrence rate of scar healing and relieve the deficiency of skin source.However, its survival rate is not high, and acellular allogeneic dermal scaffolds are expensive, heavy medical burden.Therefore, how to effectively repair the wound surface after surgical excision of scar is the main problem to be solved urgently.

Dermal loss is the main cause of unsatisfactory scar repair and recurrence.The previous clinical study of the research group found that the application of autologous epidermal basal cells and autologous skin graft obtained in real time during the operation could effectively improve the survival rate of skin graft in the treatment of wound surface (Brit J Surg, 2015).Furthermore, it is suggested that the application of autologous scar dermal scaffolds can achieve the control of skin damage in the skin harvesting area and the orthotopic transplantation of autologous scar tissue dermal scaffolds, which can effectively reduce the economic burden of patients.Therefore, the researchers wondered whether the construction of tissue-engineered skin orthotopic transplantation with autologous epidermal basal cells and autologous scar dermal scaffold combined with autologous scar dermal scaffolds to repair the wound after scar resection could improve the survival rate of skin graft and reduce scar recurrence.To this end, we plan to carry out multi-center, prospective, randomized, controlled clinical trials, aiming at proposing more effective surgical treatment guidelines for the repair of hypertrophic scar, improving the survival rate of composite skin graft, and solving the current clinical problems of hypertrophic scar repair.

ELIGIBILITY:
Inclusion Criteria:

The patient is diagnosed as hypertrophic scar and needs surgical repair; The scar size was 10cm2 to 200cm2, and the site was not limited; Patients with stable vital signs and tolerable operation indicated by routine examination; Patients in good mental state, can follow the doctor's advice, regular return; Those whom the researchers considered unsuitable for inclusion; Patients have participated in this study at any time in the past; Those whom the researchers considered unsuitable for inclusion; Patients have participated in this study at any time in the past.

Exclusion Criteria:

Those who did not meet the inclusion criteria were found after the selected subjects; The follow-up time after inclusion was less than 2 times, and the objective efficacy could not be evaluated (but the adverse reactions could be evaluated); Subjects who violate protocol requirements.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
healing rate | postsurgery week 4
  the percentage of subjects that achieved complete wound closure,complete wound closure is defined as skin conplete reepithelialization without drainage or dressing requirements.

SECONDARY OUTCOMES:
wound reducing rate | postsurgery week 4
  the rate of wound reducing based on week 4 after surgery

OTHER OUTCOMES:
recrrence rate | postsurgery month 6
  the incidence of ulcer recurrence at postsurgery month 6

CONTACTS AND LOCATIONS:
Overall Officials: ZHU JIAYUAN, Study Director — Professor, chief physician
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT04389164/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT04389164/ICF_001.pdf